CLINICAL TRIAL: NCT03517696
Title: Membrane Sweeping in Early Labor and Delivery Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study IRB approval expired
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00153394
Record Dates: First submitted 2018-04-18; First posted 2018-05-07 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-07

CONDITIONS: Early Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Intervention Model Description: Non-blinded Randomized Controlled Trial
Masking Description: Intervention is not able to be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Membrane Sweeping (Active Comparator): Membrane sweeping
  Interventions: Procedure: Membrane sweeping
- Control (No Intervention): Routine vaginal exam

INTERVENTIONS:
Procedure: Membrane sweeping — Participants assigned to membrane sweeping will have an additional exam during their initial evaluation in which the membranes will be separated from the cervix and lower part of the uterus with a finger inserted into the cervical os. This would be done with at least one rotation counterclockwise and one rotation clockwise.
  Arms: Membrane Sweeping

SUMMARY:
Membrane sweeping is a routine procedure in obstetrics in term patients. It has been shown to be effective in decreasing post term gestation and in increasing rate of spontaneous vaginal delivery when used in setting of induction of labor in nulliparous patients. The goal of this study is to determine if membranes sweeping in early labor is effective in improving delivery outcomes including decreasing rate of cesarean section.

DETAILED DESCRIPTION:
This is a non-blinded randomized controlled trial. Participants will be recruited at time of presentation to triage for labor evaluation after cervical exam. Patients with a term, singleton pregnancy who present with regular, painful contractions and a Bishop score < 7 will be recruited to the study. A random number generator will be used to create a list of random binary numbers. If the patient agrees to the study, the random number list will be used to assign the participant to membrane sweeping or no membrane sweeping. Participants assigned to membrane sweeping will have an additional exam during their initial evaluation in which the membranes will be separated from the cervix and lower part of the uterus with a finger inserted into the cervical os. This would be done with at least one rotation counterclockwise and one rotation clockwise. Those not assigned to membrane sweeping will not have an additional exam. Patients will then be managed as per their primary Obstetrics (OB) provider with the exception of no further membrane sweeping throughout the labor course.

Participants are only required to participate during initial evaluation and randomization. No extra study visits are required.

Due to the nature of the intervention, which requires a provider to perform a procedure, blinding will not be possible for this trial.

No therapy will be withheld for any patients. Their labor course will be managed as per their primary provider using standards of care.

Non-treatment group is necessary in order to exam the difference of effects between membrane sweeping and no membrane sweeping.

Patients will be removed from the study if they chose to withdraw their participation.

Participants will resume care as normal regardless of withdrawing study participation.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy at or after 39 weeks gestation, intact membranes, cephalic presentation, nulliparous, Bishop score <7, English or Spanish speaking

Exclusion Criteria:

* Prior uterine surgery precluding vaginal delivery, maternal condition precluding vaginal delivery, fetal anomaly, prior membrane stripping

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Decrease in Cesarean delivery rate | Up to 3 weeks
  Decrease in Cesarean delivery rate

SECONDARY OUTCOMES:
Time to delivery | Up to 3 weeks
  Length of labor from randomization to delivery
Operative vaginal delivery rate | Up to 3 weeks
  Assess a decrease in operative vaginal delivery
Labor augmentation rate reduction | Up to 3 weeks
  Assess the reduction in the rate of labor augmentation ( via the use of oxytocin and/or amniotomy)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne S Sheffield, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spong CY, Berghella V, Wenstrom KD, Mercer BM, Saade GR. Preventing the first cesarean delivery: summary of a joint Eunice Kennedy Shriver National Institute of Child Health and Human Development, Society for Maternal-Fetal Medicine, and American College of Obstetricians and Gynecologists Workshop. Obstet Gynecol. 2012 Nov;120(5):1181-93. doi: 10.1097/aog.0b013e3182704880. PMID 23090537
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Berghella V, Baxter JK, Chauhan SP. Evidence-based labor and delivery management. Am J Obstet Gynecol. 2008 Nov;199(5):445-54. doi: 10.1016/j.ajog.2008.06.093. PMID 18984077
- [Background] Boulvain M, Stan C, Irion O. Membrane sweeping for induction of labour. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD000451. doi: 10.1002/14651858.CD000451.pub2. PMID 15674873
- [Background] Foong LC, Vanaja K, Tan G, Chua S. Membrane sweeping in conjunction with labor induction. Obstet Gynecol. 2000 Oct;96(4):539-42. doi: 10.1016/s0029-7844(00)00995-9. PMID 11004355
- [Background] Tan PC, Jacob R, Omar SZ. Membrane sweeping at initiation of formal labor induction: a randomized controlled trial. Obstet Gynecol. 2006 Mar;107(3):569-77. doi: 10.1097/01.AOG.0000200094.89388.70. PMID 16507926
- [Background] Al-Harmi J, Chibber R, Fouda M, Mohammed ZK, El-Saleh E, Tasneem A. Is membrane sweeping beneficial at the initiation of labor induction? J Matern Fetal Neonatal Med. 2015 Jul;28(10):1214-8. doi: 10.3109/14767058.2014.947951. Epub 2014 Aug 18. PMID 25082072
- [Background] Chanrachakul B, Suthutvoravut S, Sangthawan M, Herabutya Y. Effect of lower uterine segment sweeping on progress of labor in nullipara. J Med Assoc Thai. 2001 Nov;84(11):1582-6. PMID 11853301